CLINICAL TRIAL: NCT04806399
Title: Improving Utilization of Lung Cancer Screening in Underserved PA Populations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Cure 16
Record Dates: First submitted 2021-01-08; First posted 2021-03-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: Screening Utilization
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected for assignment to the Outreach Contact with Decision Counseling Group or randomly selected for assignment to a Usual Care Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Control Group (No Intervention)
- Outreach Contact with Decision Counseling Group (Active Comparator)
  Interventions: Other: Educational Materials and Decision Counseling

INTERVENTIONS:
Other: Educational Materials and Decision Counseling — Participants in the active comparator arm will receive an introductory letter and lung cancer screening educational materials. A site care coordinator will contact each participant post receiving materials.
  Arms: Outreach Contact with Decision Counseling Group

SUMMARY:
This study is an interventional study intended to assess the impact of a centralized outreach intervention that includes shared decision-making about lung cancer screening (LCS) in LCS-eligible primary care patients. The study's goal is to increase LCS rates compared to usual care and thus reduce lung cancer deaths.

DETAILED DESCRIPTION:
The research team will select primary care practices included in areas where lung cancer mortality is high. An outreach registry of primary care patients obtaining care at participating practices who meet study eligibility criteria will be created from the electronic medical record. 500 primary care patients will be randomly selected for the Outreach Contact with Decision Counseling (OCDC) Group from this outreach registry. Patients targeted for inclusion in the study will have a scheduled primary care appointment 18-23 days after initial outreach contact.

ELIGIBILITY:
Inclusion Criteria:

* Have an upcoming office visit with a primary care physician in one of the study practices
* Between the ages of 50 and 77 (inclusive)
* History of smoking (current or former) in the electronic medical record (EMR)

Exclusion Criteria:

* Chest CT performed in the last 10 months before study initiation according to EMR
* Diagnosis of lung cancer indicated in the problem list in the EMR
* Current cancer treatment or other qualifying diagnoses that would make outreach inappropriate (e.g., dementia, hearing disability)

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Assess impact of a centralized outreach intervention that includes shared decision-making (SDM) on lung cancer screening rates compared to usual care. | 24 months
  Implement a centralized outreach intervention that includes shared decision-making (SDM) about lung cancer screening (LCS) (screening eligibility assessment, education, and decision support) in LCS-eligible primary care patients. The study's ultimate goal is to increase LCS rates compared to usual care and thus reduce lung cancer deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Etta Pisano, MD, Principal Investigator — American College of Radiology; Ronald Myers, PhD, Study Chair — Jefferson Health System
Locations (2):
- United States (2):
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Jefferson Health System, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No